CLINICAL TRIAL: NCT01884792
Title: Acute Effects of Standing on Glycemia in Prediabetic Adults: A Pilot Study
Brief Title: Effects of Standing on Glycemia in Prediabetic Adults
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Minnesota (Other)
Collaborators: Mayo Clinic (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: 1208M18741
Record Dates: First submitted 2013-06-19; First posted 2013-06-24 (Estimated); Last update posted 2014-09-15 (Estimated); Status verified 2014-09

CONDITIONS: Prediabetes
Keywords: prediabetes; physical inactivity; sedentary; standing
MeSH Terms: conditions — Prediabetic State; Sedentary Behavior

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- Sitting Oral Glucose Tolerance Test (Placebo Comparator): An OGTT is performed while the subject sits at their desk for the entire 2-hour period. 5 blood sugar measurements are taken and a 75g dextrose beverage is consumed following the first, baseline blood sugar reading. The blood sugar is then measured every 30 minutes up to 120 min.
  Interventions: Other: Sitting OGTT; Other: Standing OGTT
- Standing Oral Glucose Tolerance Test (Experimental): The participant stands at their desk for the duration of the 2-hour blood sugar test. The same procedure is performed as in the sitting condition.
  Interventions: Other: Sitting OGTT; Other: Standing OGTT
- Sitting Continuous Glucose Monitor (Placebo Comparator): A continuous blood glucose monitor is worn for 5 days while at work. In the sitting condition the participant only sits at their desk for the duration of the week. Blood sugar is monitored 4 times per day to calibrate the CGM and an accelerometer is worn to track physical activity.
  Interventions: Other: Sitting CGM; Other: Standing CGM
- Standing Continuous Glucose Monitor (Experimental): Participants are instructed to stand intermittently for at least half of their work day during this 5 day period. Blood sugar is monitored and physical activity is tracked with an accelerometer.
  Interventions: Other: Sitting CGM; Other: Standing CGM

INTERVENTIONS:
Other: Sitting OGTT
  Arms: Sitting Oral Glucose Tolerance Test; Standing Oral Glucose Tolerance Test
Other: Standing OGTT
  Arms: Sitting Oral Glucose Tolerance Test; Standing Oral Glucose Tolerance Test
Other: Sitting CGM
  Arms: Sitting Continuous Glucose Monitor; Standing Continuous Glucose Monitor
Other: Standing CGM
  Arms: Sitting Continuous Glucose Monitor; Standing Continuous Glucose Monitor

SUMMARY:
The study is a crossover, pilot trial examining the acute effects of standing on blood sugar in prediabetic, working adults. Participants will complete oral glucose tolerance testing, once while sitting and once while standing. They will also wear a continuous blood sugar monitor once while sitting at their desk for a week and once while using their desk as a sit-stand desk with a goal of standing intermittently for at least half of the work day. Physical activity levels will be measured with an accelerometer. The primary study hypothesis is that blood sugar will differ between the sitting and standing conditions for each of the tests performed.

ELIGIBILITY:
Inclusion Criteria:

* Fasting blood glucose >100 mg/dl
* Employed full-time working at least 35 hours/week
* Able to safely begin a light physical activity program

Exclusion Criteria:

* Heart disease
* Renal disease
* Peripheral neuropathy
* Retinopathy
* PAD
* Lower limb amputation
* pregnancy
* active substance abuse
* current smoker
* psychiatric disorder
* severe visual impairment
* immune-compromised individuals,
* enrollment in a physical activity study
* use of insulin or an insulin pump

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2013-03; Primary Completion 2013-07 (Actual); Study Completion 2013-09 (Actual)

PRIMARY OUTCOMES:
Blood sugar area under the curve | 2 hours
  The area under the curve following the 2 hour blood sugar tests.

SECONDARY OUTCOMES:
Accelerometer counts | 4 hours and 2 5 day periods
  Accelerometer counts in the 4 testing conditions.

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Human Services, Saint Paul, Minnesota, United States